CLINICAL TRIAL: NCT07291284
Title: A Randomized, Double-blind, Placebo-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of LP-003 Injection in Patients With Moderate to Severe Seasonal Allergic Rhinitis Inadequately Controlled by Standard-of-care
Brief Title: Efficacy and Safety of LP-003 Injection in Patients With Moderate to Severe Seasonal Allergic Rhinitis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Longbio Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P10-LP003-04
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: LP-003 (Experimental): Participants received subcutaneous of LP-003 Injection at a dose of 100 mg once every 4 weeks.
  Interventions: Biological: LP-003
- Placebo Comparator：Placebo (Placebo Comparator): Participants received subcutaneous of Placebo Injection once every 4 weeks.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: LP-003 — Participants were administered LP-003 via subcutaneous injection every 4 weeks.
  Arms: Experimental: LP-003
Biological: Placebo — Participants were administered Placebo via subcutaneous injection every 4 weeks
  Arms: Placebo Comparator：Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled phase III clinical study to evaluate the efficacy and safety of LP-003 injection in patients with moderate to severe seasonal allergic rhinitis inadequately controlled by standard-of-care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 65 years
* Subjects with SAR for at least 2 years
* At least one serum-specific IgE test for an allergen associated with the onset of allergic rhinitis during the current season or the same period
* Subjects who did not achieve satisfactory efficacy from Standard-of-Care prior to screening
* Subjects who experienced nasal symptoms for ≥ 2 days, or nasal and ocular symptoms for ≥ 1 day; with rTNSS ≥ 1 prior to randomization

Exclusion Criteria:

* Combined with non-allergic rhinitis, such as drug-induced rhinitis, vasomotor rhinitis, non-allergic rhinitis with eosinophilia syndrome, a history of acute or chronic sinusitis
* Subjects with perennial allergic rhinitis (PAR)
* Underwent any nasal or sinus surgery within 1 year prior to screening
* Presence of glaucoma, cataract, ocular herpes simplex, infectious conjunctivitis, or other ocular infections
* Clinically significant conditions upon the judgement of investigator
* Subjects with concomitant asthma who, upon the judgement of investigator, require inhaled corticosteroid treatment during the study
* The laboratory results at screening: a) white blood cell (WBC) < 2.5×10^9/L; b) aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.0 ×upper limit of normal (ULN) or total bilirubin > 1.5 ×ULN; c) Serum creatinine (Cr) > 1.5 × ULN
* Received treatment with similar drugs (e.g., Omalizumab) or used LP-003 Injection within 6 months prior to screening
* Received systemic glucocorticoids within 4 weeks prior to screening
* Received intranasal glucocorticoids, mast cell membrane stabilizers, tricyclic antidepressants, leukotriene receptor antagonists, or antihistamine medications within 1 week prior to randomization
* Received traditional Chinese medicine treatment for allergic rhinitis within the 7 days prior to randomization
* Received allergen immunotherapy within 6 months prior to screening (for those who have not completed the therapy), or within 3 years prior to screening (for those who have completed the therapy)
* Subjects for whom exposure to allergens in the home or work environment are expected to undergo significant changes during the trial, as assessed by the investigator, which may interfere with the evaluation of efficacy
* Subjects planning to travel outside their area of residence during the trial to an area without pathogenic pollen, for either 2 consecutive days or a total duration exceeding three days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean daily reflective total nasal symptom score (rTNSS) during the pollen peak period (PPP) | Up to 4 Months
  The rTNSS is a patient self-reported questionnaire of four nasal symptoms: nasal itching, nasal congestion, sneezing and rhinorrhea. Patients will report their symptoms reflected or felt over the last 12 hours. Each symptom is scored on a 0-3 scale (0 = no symptoms, 1 = mild, 2 = moderate, 3 = severe). The total score is the sum of the four items, ranging from 0 to 12, with higher scores indicating greater symptom severity.

SECONDARY OUTCOMES:
Mean daily rTNSS during the pollen period (PP) | Up to 4 Months
Mean daily instantaneous total nasal symptom score (iTNSS) during the PPP | Up to 4 Months
Mean daily iTNSS during the PP | Up to 4 Months
Mean daily rTNSS combined with rescue medication score (DNSMS) during the PPP | Up to 4 Months
  Integrates daily rTNSS (4 nasal symptoms, 0-3 each, total 0-12) and rescue medication score (0 for no rescue use and 1 for rescue use).
Mean daily total ocular symptom score (TOSS) during the PPP | Up to 4 Months
  It is derived from 2 individual ocular symptoms (itching/burning/redness, and tearing/watering), and each symptom is scored on a 0-3 scale. The daily TOSS is the sum of the two items, ranging from 0 (no symptoms) to 6 (maximum severity) per day.
Mean daily TOSS combined with rescue medication score (DNOMS) during the PPP | Up to 4 Months
  Integrates daily TOSS (2 individual ocular symptoms, 0-3 each, total 0-6) and rescue medication score (0 for no rescue use and 1 for rescue use).
Mean daily rescue medication score (RMS) during the PPP | Up to 4 Months
  The RSM is assessed based on the usage of montelukast sodium tablets, with a scoring rule of 0 points for no use and 1 point for use on the day. The mean daily RSM during the PPP is calculated as the sum of the cumulative RSM during the PPP divided by the number of days in the PPP.
Incidence of adverse events (AEs) | Up to Week 28

CONTACTS AND LOCATIONS:
Overall Officials: Xueyan Wang, Principal Investigator — Beijing Shijitan Hospital, Capital Medical University (the formerly Beijing Railway General Hospital)
Locations (1):
- Beijing Shijitan Hospital, Capital Medical University (the formerly Beijing Railway General Hospital), Beijing, China